CLINICAL TRIAL: NCT03665350
Title: Management of the Patient With Heart Failure and Diabetes: May Insulin be a Problem? A Pilot Randomized Clinical Study (Insulin-HF)
Brief Title: Insulin Treatment in Diabetic Older People With Heart Failure.
Acronym: Insulin-HF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insulin-HF study was prematurely ended due principally to low recruitment rate.
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRFMN-7468; 2018-001057-26 (EudraCT Number)
Record Dates: First submitted 2018-07-26; First posted 2018-09-11 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Heart Failure; Diabetes Mellitus, Type 2
Keywords: Heart Failure; Type 2 diabetes mellitus; Insulin; Older adults
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Intervention Model Description: The primary endpoint, glucose variability, will be computed from 3 daily glucose profiles performed before the baseline, 1, 6, 12 mo follow-up and at end study visit and calculated as the average of the three daily standard deviations. Blood glucose values will be reported by the patient in an ad hoc form and the responsible physician will input this data in the e-CRF.
  An intensive ambulatory self-monitoring of weekly body weight and possible changes in diuretic treatment is required.
  At 1, 6, 12 mo of follow up and/or at end of study visit:
  1. patients will be examined,
  2. the information about clinical events will be collected.
  3. natriuretic peptide plasma concentration, HbA1c and urinary albumin excretion will be measured Echocardiographic evaluation will be done at baseline, 1 and 12 mo after randomization.
  Central randomization in a 1:1 ratio will be performed by a web-based system.
Who Masked: Outcomes Assessor
Masking Description: Insulin-HF is a randomized, open-label, controlled, multicenter (PROBE design, prospective Randomized Open Trial with Blinded Evaluation of Outcomes), and central adjudication of adverse events.
  All study events, clinical and laboratory, will be independently validated by an Event Committee
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non insulin (No Intervention): standard care + antidiabetic therapy non insulin
- Insulin (Experimental): standard care including insulin
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Insulin as well as oral anti-diabetic drugs will be prescribed by the responsible physician and/or the diabetologist from each participating site, in conformity with the current guidelines, and the therapeutic target chosen according to patient characteristics.
  The choice of anti-diabetic medications should be guided by medical needs of each patient and taking into consideration their general safety profile.
  Arms: Insulin

SUMMARY:
Cardiac failure (HF) and type 2 diabetes mellitus (T2DM) are two clinical conditions with a significant impact on public health worldwide. In the elderly population the prevalence of T2DM is constantly increasing as well as its incidence in all Western countries including Italy. The combination of HF and T2DM is frequent and leads to an increased risk of death and of non-fatal adverse cardiovascular (CV) events which justifies the frailty of this population. Although diabetic patients (pts) with HF respond to recommended treatments for HF, the effective and safe control of blood glucose levels is still an outstanding clinical problem, since glucose lowering drugs may increase the risk of CV adverse events. Insulin, used in about 30% of diabetic patients with HF, causes adverse effects such as fluid and sodium retention and unwanted effects of hypoglycemia. Even if insulin remains a milestone in glucose lowering therapy of T2DM, its risk/benefit ratio is still controversial, more so when given to old patients with HF. The issue has gained relevance since new antidiabetic agents, as the sodium glucose co-transporter 2 (SGLT- 2) inhibitors and glucagon-like peptide (GLP-1) analogues, with a safer CV profile have been made available. While the transferability of the CV benefits attributed to the new drugs needs to be assessed in clinical practice, the present study explore the benefit/risk profile of insulin in HF.

Objectives: to assess comparatively in patients with heart failure and T2DM the benefit/risk profile over 1-year follow-up of two antidiabetic strategies, standard care with vs without insulin in terms of humoral and clinical endpoints including body weight change, all-cause mortality and burden of care components (hospitalizations for CV events and episodes of severe hypoglycemia).

DETAILED DESCRIPTION:
The project will consist in a controlled, randomized, open-label (PROBE design) multicenter, pilot study. Central randomization stratified by center, performed online, will allow a comparison of two groups of patients one receiving standard care including insulin, the other standard care without insulin. Patients considered not eligible for randomization will be included in a registry.

The first objective of this exploratory randomized study is to assess in patients with heart failure and T2DM if a standard anti-diabetic strategy which includes insulin has a different safety and efficacy profile than one without insulin. The number of patients to be included in this exploratory pilot study will be insufficient to prove or disprove a statistically significant beneficial effect of the two antidiabetic strategies on clinical events. Special care will be paid to the biologic consistency of the different endpoints, primary and secondary, even if none of them will individually yield statistically significant differences.

ELIGIBILITY:
Inclusion Criteria:

1. men and women aged ≥70 years;
2. at discharge after admission to hospital for worsening of HF or ambulatory patients with chronic HF;
3. New York Heart Association (NYHA) class II or III
4. with any level of left ventricular ejection fraction;
5. plasma natriuretic peptide (BNP) ≥200 pg/mL or N-terminal pro-BNP ≥900 pg/mL (NT pro-BNP)
6. prior history or newly diagnosed T2DM;
7. candidate by the responsible physician to insulin therapy;
8. signed informed consent.

Exclusion Criteria:

1. significant renal insufficiency (GFR <30 mL/min/1.73 m2) or severe liver disease (liver function test abnormalities (alanine or aspartate aminotransferase ≥ 3 × upper limit of normal [ULN]);
2. levels of hemoglobin <10 g/dl;
3. HbA1c ≤5% or ≥11%;
4. unstable diabetes: type of diabetes presentation in patients with an anamnesis of frequent episodes of hypoglycemia, hyperglycemic hyperosmolar state, ketoacidosis or lactic acidosis;
5. planned CV surgery or angioplasty in 3 months;
6. any non-cardiac disease that shortens life expectancy to<1 year (e.g.most cancers);
7. inability to comply with study protocol;
8. participation to another interventional clinical study.

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose variability | baseline to 12 months.
  Mean change from baseline to 12 months in glucose variability. Glucose variability is estimated as standard deviation (SD) of serial glycemic values, and is based on 3 daily glucose profiles (each with at least 5 self-measurements of blood glucose).

SECONDARY OUTCOMES:
Number of patients with episodes of hypoglycemia. | baseline, 1, 6, 12 months.
  Hypoglycemic episodes: an event accompanied or not accompanied by typical symptoms but with a measured plasma glucose concentration ≤70 mg/dl (3.9 mmol/l).
Change in body weight. | baseline, 1, 6, 12 months.
  Weight will be measured in Kg. An increase in body weight ≥2 kg gain in one week will be considered a marker of fluid congestion.
Change in plasma concentration of a natriuretic peptide | baseline, 1, 6, 12 months.
  BNP or NT-proBNP concentrations will be measured as ng/L of plasma.
Changes in urinary albumin excretion | baseline, 1, 6, 12 months.
  Urinary albumin concentration will be expressed as the urinary albumin-to-creatinine ratio (UACR), measured in milligrams per grams of creatinine, with a limit of detection of 1.5 mg/g.
Change in New York Heart Association (NYHA) class | baseline, 1, 6, 12 months.
  Any change in NYHA class. The New York Heart Association (NYHA) Functional Classification places patients in one of four categories (I through IV) based on heart failure symptoms and functional limitations. Higher NYHA classes indicate a greater heart failure severity and poorer outcome."
All-cause hospitalizations | baseline to 12 months
  Number of patients admitted to hospital for any cause.
Hospitalizations for worsening of HF. | baseline to 12 months
  Number of patients admitted to hospital for worsening of HF.
All-cause mortality | baseline to 12 months
  Number of patients who died for cardiovascular and non-cardiovascular causes.
Number of patients with episodes of ketoacidosis as evaluation of safety. | baseline to 12 months
  Ketoacidosis is defined as the presence of at least two of the following factors: a) elevated plasma glucose (>250 mg/dL), b) ketones in serum or urine and c) acidosis (serum bicarbonate <18 mEq/L and/or pH <7.30).
Number of patients with episodes of lactic acidosis as evaluation of safety. | baseline to 12 months
  Lactic acidosis is characterized by persistently increased blood lactate levels (usually >5 mmol/L) in association with metabolic acidosis.
Changes in left ventricular ejection fraction (LVEF). | baseline, 1, 6, 12 months.
  LVEF will be calculated from left ventricular volume in diastole and systole estimated by echocardiography. LVEF will be measured as percentage. A decrease in LVEF will be taken as a marker of worsening of cardiac function.
Changes in E/e'. | baseline, 1, 6, 12 months.
  E/e' ratio will be calculated from echo-Doppler recordings. As a ratio it will not have a unit of measure.
Changes in Hemoglobin A1c (HbA1c). | baseline, 1, 6, 12 months.
  HbA1c will be measured as percentage of total hemoglobin concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Staszewsky, MD, Principal Investigator — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (3):
- Italy (3):
  - Ospedale Bolognini di Seriate, Seriate, BG
  - Ospedale Treviglio, Treviglio, BG
  - Ospedale di Passirana, Passirana, MI

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Diabetes Association. 11. Older Adults: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018 Jan;41(Suppl 1):S119-S125. doi: 10.2337/dc18-S011. PMID 29222382
- [Background] Aspromonte N, Gulizia MM, Di Lenarda A, Mortara A, Battistoni I, De Maria R, Gabriele M, Iacoviello M, Navazio A, Pini D, Di Tano G, Marini M, Ricci RP, Alunni G, Radini D, Metra M, Romeo F. ANMCO/SIC Consensus Document: cardiology networks for outpatient heart failure care. Eur Heart J Suppl. 2017 May;19(Suppl D):D89-D101. doi: 10.1093/eurheartj/sux009. Epub 2017 May 2. PMID 28751837
- [Background] Bozkurt B, Aguilar D, Deswal A, Dunbar SB, Francis GS, Horwich T, Jessup M, Kosiborod M, Pritchett AM, Ramasubbu K, Rosendorff C, Yancy C; American Heart Association Heart Failure and Transplantation Committee of the Council on Clinical Cardiology; Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular and Stroke Nursing; Council on Hypertension; and Council on Quality and Outcomes Research. Contributory Risk and Management of Comorbidities of Hypertension, Obesity, Diabetes Mellitus, Hyperlipidemia, and Metabolic Syndrome in Chronic Heart Failure: A Scientific Statement From the American Heart Association. Circulation. 2016 Dec 6;134(23):e535-e578. doi: 10.1161/CIR.0000000000000450. Epub 2016 Oct 31. No abstract available. PMID 27799274
- [Background] Cosmi F, Shen L, Magnoli M, Abraham WT, Anand IS, Cleland JG, Cohn JN, Cosmi D, De Berardis G, Dickstein K, Franzosi MG, Gullestad L, Jhund PS, Kjekshus J, Kober L, Lepore V, Lucisano G, Maggioni AP, Masson S, McMurray JJV, Nicolucci A, Petrarolo V, Robusto F, Staszewsky L, Tavazzi L, Teli R, Tognoni G, Wikstrand J, Latini R. Treatment with insulin is associated with worse outcome in patients with chronic heart failure and diabetes. Eur J Heart Fail. 2018 May;20(5):888-895. doi: 10.1002/ejhf.1146. Epub 2018 Feb 28. PMID 29488676
- [Background] DeVries JH. Glucose variability: where it is important and how to measure it. Diabetes. 2013 May;62(5):1405-8. doi: 10.2337/db12-1610. PMID 23613566
- [Background] DeFronzo RA, Cooke CR, Andres R, Faloona GR, Davis PJ. The effect of insulin on renal handling of sodium, potassium, calcium, and phosphate in man. J Clin Invest. 1975 Apr;55(4):845-55. doi: 10.1172/JCI107996. PMID 1120786
- [Background] Giorda CB, Rossi MC, Ozzello O, Gentile S, Aglialoro A, Chiambretti A, Baccetti F, Gentile FM, Romeo F, Lucisano G, Nicolucci A; HYPOS-1 Study Group of AMD. Healthcare resource use, direct and indirect costs of hypoglycemia in type 1 and type 2 diabetes, and nationwide projections. Results of the HYPOS-1 study. Nutr Metab Cardiovasc Dis. 2017 Mar;27(3):209-216. doi: 10.1016/j.numecd.2016.10.005. Epub 2016 Nov 18. PMID 28017523
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Colvin MM, Drazner MH, Filippatos GS, Fonarow GC, Givertz MM, Hollenberg SM, Lindenfeld J, Masoudi FA, McBride PE, Peterson PN, Stevenson LW, Westlake C. 2017 ACC/AHA/HFSA Focused Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. Circulation. 2017 Aug 8;136(6):e137-e161. doi: 10.1161/CIR.0000000000000509. Epub 2017 Apr 28. No abstract available. PMID 28455343
- [Background] ORIGIN Trial Investigators; Gerstein HC, Bosch J, Dagenais GR, Diaz R, Jung H, Maggioni AP, Pogue J, Probstfield J, Ramachandran A, Riddle MC, Ryden LE, Yusuf S. Basal insulin and cardiovascular and other outcomes in dysglycemia. N Engl J Med. 2012 Jul 26;367(4):319-28. doi: 10.1056/NEJMoa1203858. Epub 2012 Jun 11. PMID 22686416